CLINICAL TRIAL: NCT00531544
Title: A SU011248 Expanded Access Protocol for Metastatic RCC Patients Who Are Ineligible for Participation in Other SU011248 Protocols But May Derive Benefit From Treatment With SU011248
Brief Title: A SU011248 Expanded Access Protocol for Systemic Therapy of Patients With Metastatic Renal Cell Carcinoma Who Are Ineligible for Participation in Other SU011248 Protocols But May Derive Benefit From Treatment With SU011248
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAC#2061 043
Record Dates: First submitted 2007-09-17; First posted 2007-09-19 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: SU011248 — SU011248 Expanded Access Protocol for Systemic Therapy

SUMMARY:
A SU011248 expanded access protocol for systemic therapy of patients with metastatic Renal Cell Carcinoma who are ineligible for participation in other SU011248 protocols but may derive benefit from treatment with SU011248

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic Renal Cell Carcinoma who are ineligible for participation in other SU011248 protocols but may derive benefit from treatment with SU011248

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2007-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Efficacy | 2001-2012

CONTACTS AND LOCATIONS:
Overall Officials: Shouki Bazarbashi, MD, Principal Investigator — KFSH&RC, Riyadh, Saudi Arabia
Locations (1):
- KFSH&RC, Riyadh, Saudi Arabia